CLINICAL TRIAL: NCT06315465
Title: Efficacy of Modified Atkin's Diet as add-on Therapy in Comparison With Standard of Care in Children With Autism Spectrum Disorder A Randomized Controlled Trial
Brief Title: Efficacy of MAD as add-on Therapy in Comparison With Standard of Care in Children With ASD
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMSA00647
Record Dates: First submitted 2024-02-29; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Modified Atkins Diet; Autism Spectrum Disorder; Standard of Care
Keywords: Modified Atkin's Diet; Autism Spectrum Disorder; Standard of care
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open Label Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Atkin's diet with standard of care arm (Experimental): Group I will receive Modified Atkin's Diet with standard of care whereas Group II will receive standard of care alone. Children randomized into Group I, initial workup for Modified Atkin's Diet will be done in the form of Electrocardiogram, Renal Function Tests, Liver Function Tests, Complete Blood Counts, Lipid profile, Urine calcium creatinine ratio and Ultrasound Pelvis for nephrocalcinosis. If pre KD work up is normal, then Modified Atkin's Diet will be initiated in the ratio of 1:1.Urine ketones will be checked daily using ketone dipsticks. Telephonic contacts will be made in regular intervals every week to further ensure compliance at home, and to ensure proper understanding and confidence of parents. Those children who are unable to tolerate taking adequate ketogenic diet therapy requiring discontinuation of therapy, will be considered as deviates. First follow-up will be at 4 weeks of treatment initiation, followed by at 8, 12, 16, 20 and 24 weeks.
  Interventions: Dietary Supplement: Modified Atkin's Diet with standard of care; Other: Standard of Care
- Standard of care arm (Other): * Standard of care intervention plan will be devised for each subject based on the principles of -
  * Behavioral therapy
    1. Behavioral modification techniques
    2. Psycho education
    3. Cognitive behavioral therapy
    4. Activity based interventions like eye contact exercises, attention enhancement exercises, self-help skills
    5. Speech therapy
    6. Parental training
  * Occupational therapy
  * Sensory integration therapy
  * Pharmacotherapy - Anti-psychotic medications
  * The parents of the children will be called telephonically every weekly to check for any issues and reinforcement to ensure appropriate regular behavioural intervention to be provided to the child.
  * Physical follow up - 4, 8, 12, 16, 20, 24 weeks
  * Follow up assessments - 12 weeks (3 months) & 24 weeks (6 months)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Modified Atkin's Diet with standard of care — children who have given their consent and are randomized into Group I arm receives Modified Atkins Diet along with standard of care after completion of baseline investigations. Modified Atkin's Diet will be started in ratio of 1:1 and compliance is monitored by urine ketones. Followup will be done telephonically to check for compliance , adverse events at every 4 week intervals till 24 weeks.
  Arms: Modified Atkin's diet with standard of care arm
Other: Standard of Care — Standard of care intervention plan will be devised for each subject which includes Behavioral therapy , Psychoeducation, Activity based interventions like attention enhancement exercises, self help skills, Occupational therapy, Pharmacotherapy, Sensory integration therapy. The parents of the children will be called telephonically every weekly to check for any issues and reinforcement to ensure appropriate regular behavioral intervention to be provided to the child. Physical follow up will be done every 4 weekly till 24 weeks.

SUMMARY:
In general ketogenic diet is a recognized as an efficient non pharmacological treatment for children with refractory epilepsy. However, in the last decade, it has been tried for many neurological disorders in children including ASD, neurodegenerative disorders.

Studies have shown that KD also helps in improvement of cognition, social skills, language function, and stereotypies. There is a limited number of reports of improvements after KD treatment, was insufficient evidence to attest the practicability of the KD as a treatment for ASD, but it is still a good indicator that this diet is a promising therapeutic option for this disorder. There are no major RCT's, hence raises concerns about the reliability and generalizability of findings. Majority of studies have used combined ketogenic diet therapy rather than single diet therapy and not many studies have compared add-on dietary intervention with standard of care. When compared to classic KD diet Modified Atkin's Diet is less restrictive, more palatable, more feasible and early response can be achieved. In summary, the rationale for conducting this study lies in the importance of add on dietary therapy in form of Modified Atkin's Diet along with standard of care for improvement of behavioral symptoms in children with ASD aged 3-8 years.

This study aims to provide valuable insights that it can improve behavioral symptoms in ASD, early and ultimately improve the developmental outcomes in these children.

DETAILED DESCRIPTION:
* All the children presenting to Paediatrics OPD and Autism clinic in the Child Neurology division will be screened and those fulfilling the inclusion and exclusion criteria will be enrolled into the study
* Informed consent will be taken from parents for the study
* Baseline demographic details and following evaluation will be done -

  1. Autism severity assessment using CARS -2, ABC
  2. Neurocognitive assessment using (DQ/IQ/SQ) -VSMS
  3. Behavioral assessment using CBCL
  4. Sleep related issues using CSHQ After initial assessment children are randomized into Group I and Group II using computer generated random numbers.

Group I-Modified Atkin's Diet with standard of care arm

* Group I will receive Modified Atkin's Diet with standard of care whereas Group II will receive standard of care alone.
* Children randomized into Group I, initial workup for Modified Atkin's Diet will be done in the form of Electrocardiogram, Renal Function Tests, Liver Function Tests, Complete Blood Counts, Lipid profile, Urine calcium creatinine ratio and Ultrasound Pelvis for nephrocalcinosis. If pre KD work up is normal, then Modified Atkin's Diet will be initiated in the ratio of 1:1.
* Urine ketones will be checked daily using ketone dipsticks
* Telephonic contacts will be made in regular intervals every week to further ensure compliance at home, and to ensure proper understanding and confidence of parents
* Those children who are unable to tolerate taking adequate ketogenic diet therapy requiring discontinuation of therapy, will be considered as deviates
* First follow-up will be at 4 weeks of treatment initiation, followed by at 8, 12, 16, 20 and 24 weeks
* Compliance rate and adverse events will also be calculated from patient diary/log
* Those children who are unable to tolerate taking adequate ketogenic diet therapy requiring discontinuation of therapy, will be considered as deviates
* First follow-up will be at 4 weeks of treatment initiation, followed by at 8, 12, 16, 20 and 24 weeks
* Compliance rate and adverse events will also be calculated from patient diary/log
* Every alternate subject from each category, pre - intervention f MRI and 3 months post intervention f MRI is done (total 10 subjects) Group II -Standard of care arm
* Standard of care intervention plan will be devised for each subject based on the principles of -
* Behavioral therapy

  1. Behavioral modification techniques
  2. Psycho education
  3. Cognitive behavioral therapy
  4. Activity based interventions like eye contact exercises, attention enhancement exercises, self-help skills
  5. Speech therapy
  6. Parental training
* Occupational therapy
* Sensory integration therapy
* Pharmacotherapy - Anti-psychotic medications
* The parents of the children will be called telephonically every weekly to check for any issues and reinforcement to ensure appropriate regular behavioural intervention to be provided to the child.
* Physical follow up - 4, 8, 12, 16, 20, 24 weeks
* Follow up assessments - 12 weeks (3 months) & 24 weeks (6 months)

Functional MRI acquisition Every 4th subject from each group who provide consent for doing a f-MRI, will undergo a pre-intervention f-MRI and post-intervention f-MRI at 3 months follow-up (10 subjects in each arm, i.e. 20 subjects) These investigations would be done free of cost for the patients. The data will be compared with fMRI data of controls (retrospective data of children with dyslexia who received AI enabled-remedial intervention alone (for 6 weeks) as a part of a previous study by Dr Sayoni Roy Chowdhary, under the guidance of Prof Sheffali Gulati as Chief guide, after ethical clearance). The data will also be compared with the historical data of typical readers, acquired using the same f-MRI protocol at our center

ELIGIBILITY:
Inclusion Criteria:

* 1. Children aged 3 to 8 years diagnosed with Autism Spectrum Disorder according to DSM -V criteria

Exclusion Criteria:

1. Diagnosed genetic and metabolic syndromes
2. Pre-existing food fads
3. Associated seizure disorder/epilepsy syndrome
4. Chronic systemic illness
5. Received any form of dietary therapy in the previous 6 months
6. Not on stable standard of care therapy or changes in antipsychotic medications over the last 1 month
7. Refusal of consent

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of add-on Modified Atkin's Diet therapy with standard of care as compared to standard of care alone in children with Autism Spectrum Disorder aged 3-8 years | 3 months
  Proportion of children with minimum significant reduction of Childhood Autism Rating Scale (CARS-2) score (defined by ≥ 4.5 reduction) in both arms. Childhood Autism Rating Scale is an evaluation tool used for identifying autism and determining the severity of autism spectrum disorder. It can be used in children 2 years and older with Autism Spectrum Disorder. It contains total 15 domains and each domain have score from 0-4. Total score 15 to 60 and total score of less than 30 indicates non autism, 30-36.5 indicates mild to moderate autism, 37-60 is considered as severe autism

SECONDARY OUTCOMES:
To evaluate the efficacy of add-on Modified Atkin's Diet therapy with standard of care as compared to standard of care alone in children with Autism Spectrum Disorder aged 3-8 years | 6 months
  Proportion of children with minimum significant reduction of Childhood Autism Rating Scale (CARS-2) score (defined by ≥ 4.5 reduction) in both arms. Childhood Autism Rating Scale is an evaluation tool used for identifying autism and determining the severity of autism spectrum disorder. It can be used in children 2 years and older with Autism Spectrum Disorder. It contains total 15 domains and each domain have score from 0-4. Total score 15 to 60 and total score of less than 30 indicates non autism, 30-36.5 indicates mild to moderate autism, 37-60 is considered as severe autism
To compare the change in the cognitive ability as measured by Developmental Quotient(DQ)in children receiving Modified Atkin's Diet with standard of care vs standard of care alone in children with Autism Spectrum disorder aged 3-8 years. | 6 months
  Developmental Quotient is assessed in both arms pre and post diet therapy using Developmental profile -3 (DP-3).It utilizes input from parents or caregivers to provide scores in five areas of development: physical, adaptive behavior, social emotional , cognitive, and communication. It provide five scales each with 34 to 38 items, designed to assess the development and functioning of children from birth through age12. Scores less than 70 is considered delayed, 70-84 is considered below average,85-115 is considered average, 116-130 is considered above average and more than 130 is considered well above average.
To compare the change in the cognitive ability as measured by Social Quotient(SQ)in children receiving Modified Atkin's Diet with standard of care vs standard of care alone in children with Autism Spectrum disorder aged 3-8 years. | 6 months
  Social Quotient (SQ) is assessed in both arms pre and post therapy using Vineland Social Maturity Scale. It is generally used to determine three related but different aspects, which is 1)social and adaptive functions,2)level of disability, 3) intelligence. It contains 89 items in 8 domains and assess from 0 to 15 years. Scores of less than 70 is considered as intellectual disability, 70-79 as borderline impaired or delayed, 80-89 is considered as low average, 90-109 is considered as average,110-119 is considered as high average.
To compare the change in the cognitive ability as measured by Intelligence Quotient(IQ)in children receiving Modified Atkin's Diet with standard of care vs standard of care alone in children with Autism Spectrum disorder aged 3-8 years. | 6 months
  Intelligence Quotient (IQ)is assessed in both arms pre and post therapy using Malins Intelligence Scale for Indian children (MISC). It includes both verbal and performance scales. Total 11 subtests are used of which 6 are verbal tests and 5 are performance tests. This test yields three scores: verbal IQ, performance IQ, and full scale IQ scores. Scores of less than 70 is considered as Intellectual disability, 70-79 as borderline impaired or delayed, 80-89 is considered as low average, 90-109 is considered as average,110-119 is considered as high average.
To compare the quantitative reduction in behavioral problems using Child Behavior Checklist (CBCL) in children receiving Modified Atkin's Diet with standard of care vs standard of care alone in children with Autism Spectrum Disorder aged 3-8 years. | 6 months
  Behavior problems like inattention, hyperactivity, aggression are assessed pre and post therapy in both arms using Child Behavior Checklist. This checklist can assess behavior in the following profiles: Anxious/depressed, withdrawn, sleep problems, somatic problems, aggressive behavior, or destructive behavior. Based on these three scores are generated, Total score, Externalizing problem scale , and Internalizing problem scale. Any score that falls below the 93rd percentile is considered normal, scores between the 93-97th percentile are borderline clinical, and any score above the 97th percentile are in the clinical range.
To compare the change in sleep related problems using Children's Sleep Habit Questionnaire (CSHQ)children receiving Modified Atkin's Diet with standard of care vs standard of care alone in children with Autism Spectrum Disorder age | 6 months
  The CSHQ is a parent-rated questionnaire comprised of 45 items; 33 scored questions, and 7 additional items intended to provide other relevant information pertaining to sleep behavior (e.g., nocturnal body pains) Each scored question is rated on a 3-point scale as occurring "usually" (i.e., 5-7 times within the past week), "sometimes" (i.e., 2-4 times within the past week), or "rarely" (i.e., never or 1 time within the past week).A number of items on the questionnaire are reverse-scored, so that higher scores consistently indicate problem behaviors. Ratings are combined to form eight subscales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night wakings, Parasomnias, Sleep Disordered Breathing, and Daytime Sleepiness. A Total Sleep Disturbances score is calculated as the sum of all CSHQ scored questions, and can range from 33 to 99
To compare the resting state fMRI findings in a subset of patients in the two arms | 6 months
  To observe the changes in resting state functional MRI in both arms (pre and post therapy) at 6 months
To assess the compliance in children with Autism Spectrum Disorder receiving add-on Modified Atkin's Diet with standard of care | 6 months
  compliance will be monitored using Compliance diary
To assess the adverse effect profile in children with Autism Spectrum Disorder receiving add-on Modified Atkin's Diet with standard of care | 6 months
  adverse effects will be checked by Patient diet log

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — All India Institute of Medical Sciences